CLINICAL TRIAL: NCT03669367
Title: EFFECTS OF ABATACEPT ON THE PROGRESSION TO RHEUMATOID ARTHRITIS IN PATIENTS WITH PALINDROMIC RHEUMATISM (PALABA)
Brief Title: EFFECTS OF ABATACEPT on the Progression to Rheumatoid Arthritis(PALABA Study)
Acronym: PALABA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project manager Clinical Trial Unit, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALABA 2017-004543-20
Record Dates: First submitted 2018-07-26; First posted 2018-09-13 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2024-07

CONDITIONS: Palindromic Rheumatism, Wrist
MeSH Terms: conditions — Palindromic rheumatism | interventions — Abatacept

STUDY DESIGN:
Intervention Model Description: National multi-center study, open, controlled and randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- abatacept (Experimental): abatacept monotherapy (subcutaneous route).: 125 mg solution for injection in pre-filled syringe. In the first year (0-12 months) at a a dose of 125 mg per week (full dose) and in the second year (12-24 months) at a dose of 125 mg every other week (q2w) (optimized dose) injection) - 125 mg x week - subcutaneous use.
  Interventions: Drug: Abatacept Injection
- hydroxycloroquina (Active Comparator): Hydroxyclorquina (Coated tablet)- (5 mg/Kg/day) monotherapy for 2 years (0-48 months)
  Interventions: Drug: hydroxycloroquina

INTERVENTIONS:
Drug: Abatacept Injection — Abatacept subcutaneous in monotherapy 125 mg/week during the first year (12 months). Abtacept subcutaneus in monotherapy 125 mg/2weeks during the second year.
  Other Names: ORENCIA
  Arms: abatacept
Drug: hydroxycloroquina — oral hydroxycloroquina 5 mg/Kg/day for 2 years (0-48 months)
  Arms: hydroxycloroquina

SUMMARY:
The main objective of this trial is to test the hypothesis that abatacept can reduce the progression of rheumatoid arthritis in ACPA+ or RF+ patients with palindromic rheumatism compared with patients treated with hydroxychloroquine.

DETAILED DESCRIPTION:
The main objective of this trial is to test the hypothesis that abatacept can reduce the progression of rheumatoid arthritis in ACPA+ or RF+ patients with palindromic rheumatism compared with patients treated with hydroxychloroquine.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PR according to Guerne and Weissman modified criteria (18) and with:
* Disease evolution > 3 months and < 24 months.
* ACPA positivity proven by ELISA test or chemiluminescence (CCP2) and/or Rheumatoid factor positivity (ELISA, nephelometry or chemiluminescence).
* Greater than 18 years of age.

Exclusion Criteria:

* Persistent arthritis: (involvement in one or more joints > 1 week).
* Criteria of other rheumatic diseases (RA, SLE, etc.).
* Evidence of radiographic damage (join erosions).
* Absence of ACPA or RF.
* Contraindication or intolerance to study drugs (abatacept or hydroxychloroquine).
* Steroid treatment one month before study entry.
* Previous antitrheumatic therapy with synthetic DMARDS (methotrexate, leflunomide, sulfasalazine, cyclosporine, antimalarials.) or biological DMARDs.
* Pregnant women or who want to be pregnant during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The main objective of this trial is to test abatacept efficacy | At any time during the follow-up (up to 24 months)
  number of participants developed persistent arthritis fulfilling criteria of Rheumatoid Arthritis according to EULAR/ACR 2010 classification criteria persistent arthritis (RA criteria)

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as asesed | At any time during the follow-up (up to 24 months)
  Number of participants with treatment-related adverse events as asesed
number of participants with titles positives on serum ACPA.(anti-CarP antibodies) | At any time during the follow-up (up to 24 months)
  number of participants with titles positives on serum ACPA.(anti-CarP antibodies)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided